CLINICAL TRIAL: NCT05885334
Title: Caregivers Training Using Artificial Intelligence and Virtual Reality
Acronym: RealityCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, José Joaquín Mira Solves, Principal investigator, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TED2021-130383B-I00
Record Dates: First submitted 2023-03-31; First posted 2023-06-01 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Medication Errors and Other Product Use Errors and Issues; Caring

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Naturalistic Intervention (Placebo Comparator): Natural intervention (actual provision of information and answering of questions). This arm will evaluate the natural learning during the action.
  Interventions: Other: Control
- Virtual Reality (Experimental): Virtual Reality intervention specifically designed for this study. Using VR to learn procedures will encourage caregivers to learn in a fully immersive and participatory environment where they will have to interact with the virtual content, enhancing their learning experience.
  Interventions: Other: Virtual Reality
- Augmented Reality (Experimental): Augmented Reality Intervention specifically designed for this study. This intervention will increase participants' skills through active learning as they interact with real-world care situations while receiving simultaneous support from AR devices.
  Interventions: Other: Augmented Reality

INTERVENTIONS:
Other: Control — Caregivers will not receive any educational solution different than what is done by routine in centers. After six months, performance in caregivers tasks will be video recorded.
  Arms: Naturalistic Intervention
Other: Virtual Reality — Caregivers will receive a educational solution of virtual reality videos with care situations simulations for 1h. After six months, performance in caregivers tasks will be video recorded.
  Arms: Virtual Reality
Other: Augmented Reality — Caregivers will receive a educational solution of augmented reality videos with care situations simulations for 1h. After six months, performance in caregivers tasks will be video recorded.
  Arms: Augmented Reality

SUMMARY:
What the investigators propose. The use of disruptive digital technologies for their potential to improve caregivers training, ensure the adequacy of care and achieve a greater quality of life for recipients; increase the efficiency of interventions to support caregivers, quickly reaching a greater number of people; democratize access to adequate care; dignify the lives of people working in this sector, mostly women; develop a new sector of the economy by promoting the modernization and technification of the sector. The project seeks to place people at the center of interventions while respecting their digital rights. The investigators identify as disruptive technologies those based on recent innovations (such as virtual and augmented reality, artificial intelligence AI) with a high capacity to evolve rapidly, adapting to very different needs and sectors, and a high capacity to generate new business models. These emerging technologies open up new opportunities to improve the well-being of dependent people, provide new skills (including soft ones) to caregivers and would be also useful against gender stereotypes in the caregiving sector.

DETAILED DESCRIPTION:
Feasibility study of VR/AR/AI applications to the context of caregiver training in three phases including mixed methodologies: (1) qualitative (to collect key information to elaborate immersive environments for VR/AR-based interventions), (2) experimental (to test the effectiveness of the intervention targeting caregivers (informal and formal) to provide safe home care, including cost-effectiveness analysis, (3) prototype development to capture and analyze the performance of home care to promote improvements in training programs through VR/AR. General objective. The primary aim is to investigate whether the provision of care in the home of persons suffering multiple pathologies and polypharmacy by trained formal/informal caregivers using VR/AR is more efficient than traditional training. Secondary aims are to provide competencies (knowledge, skills, and attitudes) that contribute to reducing care and medication errors made by caregivers, contributing to recipients staying at home for as long as possible; and to determine to what extent AI allows us to continuously update the VR training material. This Project is in line with the WHO SDG3 "Ensure healthy lives and promote well-being for all at all ages". It also responds to the WHO challenge of Medication Without Harm. At national level, this study reinforces those policies aim to strengthen the new care economy and reduce the gender equality gap (Component 22, June 16, 2021).

ELIGIBILITY:
Study participants are qualified or unqualified caregivers who oversee patients in one of two groups: 1) multi-pathological, polymedicated, dependent, and 2) devices and catheters (oncological, ostomy, etc.). To facilitate recruitment, each centre will be provided with templates adjusted to the participants and arms to which they are committed. The inclusion criteria for each group are detailed below.

Inclusion criteria for carers of multi-pathological, polymedicated and dependent patients

* Qualified or unqualified carers caring for multi-pathological patients (coexistence of two or more chronic conditions lasting one year or more, requiring continuous medical assistance or limiting daily activities), polymedicated (simultaneous daily treatment of 5 or more drugs) and Barthel equal or lower than 55.
* Carers who are in charge of this person for at least 6 months of the year.
* Residence in C. Valenciana, Andalusia, R. de Murcia, C. Madrid and Catalonia (in the home of the patient or relative).

Inclusion criteria for caregivers of patients with devices and catheters

* Qualified or unqualified caregivers in charge of patients with a fixed catheter who require care from another person.
* Carers who are in charge of that person for at least 6 months of the year.
* Residence in C. Valenciana, Andalucía, R. de Murcia, C. Madrid and Cataluña (in the patient's or relative's home).

Exclusion criteria

The exclusion criteria are common to both groups of carers:

* Caregivers of patients who had filed a patrimonial claim in the last 5 years.
* Carers of part-time residents in nursing homes.
* Carers with a health profession.
* Carers of dependent elderly people who do not meet the inclusion criteria.
* Carers with experience in using VR or AR for a similar purpose.
* Carers over 90 years of age.
* Carers with more than two dependents.
* Carers with problems of vertigo, tinnitus, motion sickness, epilepsy, seizures or similar symptoms, severe cardiac conditions or wearing a cardiac pacemaker or hearing aid.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Change in number of caring errors and medication errors | 6 months
  The evaluation of the effectiveness of each of the arms will be measured, among other ways, by recording two attempts to execute the care situation to be trained in the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación Fisabio, Sant Joan d'Alacant, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ballester P, Gil-Hernandez E, Perez-Esteve C, Guilabert M, Carrillo I, Arroyo A, Cobos A, Mira JJ. Medication incidents and informal caregiver burden: A cross-sectional study. J Healthc Qual Res. 2025 Dec 24;41(2):101175. doi: 10.1016/j.jhqr.2025.101175. Online ahead of print. PMID 41447744
- [Derived] Mira JJ, Ballester P, Gil-Hernandez E, Sambrano Valeriano L, Alvarez Gomez E, Olier Garate C, Marquez Ruiz A, Acedo Torrecilla M, Arroyo Rodriguez A, Hidalgo Galache E, Navas Gutierrez P, Perez-Jover V, Lorenzo Martinez S, Carrillo Murcia I, Fernandez Peris C, Sanchez-Garcia A, Vicente Ripoll MA, Cobos Vargas A, Perez-Perez P, Guilabert Mora M. Safe Care and Medication Intake Provided by Caregivers at Home: Reality Care Study Protocol. Healthcare (Basel). 2023 Aug 3;11(15):2190. doi: 10.3390/healthcare11152190. PMID 37570430